CLINICAL TRIAL: NCT05494567
Title: Efficacy of Tadalafil and Solifenacin Versus Tamsulosin and Solifenacin Combination Therapy for the Treatment of Benign Prostatic Hyperplasia With Overactive Bladder: A Randomized Controlled Trial
Brief Title: Efficacy of Tadalafil/Solifenacin VS Tamsulosin/Solifenacin Combination Therapy for BPH/OAB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohammed Hegazy, principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tadalafil for BPH/OAB
Record Dates: First submitted 2022-08-07; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Benign Prostatic Hyperplasia; Overactive Bladder
Keywords: Benign Prostatic Hyperplasia; Overactive Bladder; tadalafil; combination therapy for BPH
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder, Overactive | interventions — Tadalafil; Tamsulosin; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tadalafil / solifenacin combination therapy (Active Comparator): Patients will be treated by combination of Tadalafil 5 mg + solifenacin 10 mg once daily for 12 weeks
  Interventions: Drug: Tadalafil 5mg; Drug: solifenacin 10 mg
- Tamsulosin / solifenacin combination therapy (Active Comparator): Patients will be treated by combination of Tamsulosin 0.4 mg + solifenacin 10 mg once daily for 12 weeks
  Interventions: Drug: Tamsulosin Hcl 0.4 mg; Drug: solifenacin 10 mg

INTERVENTIONS:
Drug: Tadalafil 5mg — patients with BPH/OAB will be treated with combination therapy of tadalafil plus solifenacin for 12 weeks in group 1
  Other Names: rectalis 5 mg
  Arms: Tadalafil / solifenacin combination therapy
Drug: Tamsulosin Hcl 0.4 mg — patients with BPH/OAB will be treated with combination therapy of tamsulosin plus solifenacin for 12 weeks in group 2
  Other Names: tamsulosin 0.4 mg
  Arms: Tamsulosin / solifenacin combination therapy
Drug: solifenacin 10 mg — patients with BPH/OAB will be treated with combination therapy of tadalafil plus solifenacin in group 1 and tamsulosin plus solifenacin in group 2 for 12 weeks

SUMMARY:
The investigators will compare the efficacy and safety of tadalafil/solifenacin combination therapy versus tamsulosin/solifenacin combination therapy for the treatment of BPH/OAB in a randomized controlled trial (RCT).

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is one of the most commonly diagnosed diseases in aging men worldwide. It is commonly associated with bothersome lower urinary tract symptoms (LUTS) including voiding symptoms such as decreased force of stream, intermittent stream, hesitancy and sensation of incomplete bladder emptying and storage symptoms such as frequent urination, urgency and nocturia. LUTS especially storage symptoms interfere with the daily activities and adversely affect the quality of life (QoL).

Alpha-1 adrenergic receptor blockers have been used as a first-line treatment of LUTS suggestive of BPH (LUTS/BPH). Phosphodiesterase 5 inhibitors (tadalafil) have recently been used as initial treatment of LUTS/BPH. It was confirmed that once daily use of tadalafil 5 mg as a monotherapy is safe and has similar efficacy when compared to tamsulosin.

Combination therapy could be used in patients who have BPH with overactive bladder (BPH/OAB) and still have persistent storage symptoms despite α1- adrenergic blockers. Anticholinergics in combination with α1- adrenergic blockers have been reported to be effective in those patients. Moreover, it has been reported that tadalafil has similar efficacy and safety to solifenacin when used in combination with tamsulosin for patients with persistent storage symptoms refractory to α1- adrenergic blockers. In another study, tadalafil/mirabegron combination therapy was used for BPH/OAB and its effect appeared to be greater than the effect of tadalafil monotherapy. Also, the combination therapy of tadalafil and solifenacin was approved to achieve higher response than tadalafil monotherapy in improvement of persistent storage symptoms associated with BPH.

It was established that tadalafil can be used as a monotherapy to relieve both voiding and storage LUTS and it can be used in combination with tamsulosin or mirabegron to treat BPH/OAB. However, there is limited evidence regarding the efficacy and safety of the combined use of tadalafil and solifenacin for the treatment of BPH/OAB. Therefore, in this study, the investigators will compare the efficacy and safety of tadalafil/solifenacin combination therapy versus tamsulosin/solifenacin combination therapy for the treatment of BPH/OAB in a randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent and reply to questionnaires.
2. Age ≥ 45 years
3. IPSS ≥ 8
4. OABSS ≥ 5, urgency subscore ≥2

Exclusion Criteria:

1. Untreated urinary tract infection (UTI).
2. Postvoid residual (PVR) more than 150 mL
3. Neurogenic lower urinary tract dysfunction (LUTD).
4. Depression or any psychogenic disorders.
5. Diabetes mellitus, hypertension or severe cardiovascular disease.
6. Prior radiation therapy to the pelvic area.
7. Prostate cancer or bladder tumor.
8. Past history of tuberculosis
9. Allergy or contraindication to the used medications
10. Urethral stricture
11. Indwelling urethral catheter
12. Vesical stone.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients suffering from BPH/OAB will be asked to participate in this study
Enrollment: 60 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change in international prostate symptom score (IPSS) from baseline | 3 months
  Change in IPSS from baseline will be compared. The change of -3 will be estimated as the minimal threshold for a meaningful change. The score has a range from 0 to 35 and higher scores means a worse outcome.
Change in overactive bladder symptom score (OABSS) from baseline | 3 months
  Change in OABSS from baseline will be compared. The change of -3 will be estimated as the minimal threshold for a meaningful change. The score has a range from 0 to 15 and higher scores means a worse outcome.
Change in IPSS-quality of life (QoL) score from baseline | 3 months
  Change in IPSS-QoL score from baseline will be compared. It is a single question with a score ranges from 0 to 6 and higher scores means a worse outcome.
Change in ultrasound measurement of post-void residual urine (PVR) from baseline | 3 months
  Change in PVR from baseline will be compared.
Change in maximum flow rate (Qmax) from baseline | 3 months
  Change in Qmax from baseline will be compared.
Adverse effects | 3 months
  Appearance of adverse effects related to the used medications will be reported.

SECONDARY OUTCOMES:
change in international index of erectile function-15 (IIEF-15) | 3 months
  change in IIEF-15 in sexually active patients will be compared.
change in ejaculatory domain of male sexual health questionnaire (Ej-MSHQ) | 3 months
  change in Ej-MSHQ in sexually active patients will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Hegazy, Principal Investigator — Mansoura University; Ahmed Elhefnawy, Study Director — Mansoura University
Locations (1):
- Urology and Nephrology center, Al Mansurah, Egypt